CLINICAL TRIAL: NCT02390622
Title: Fecal Microbiota Transplantation Restores Dysbiosis in Patients With Methicillin Resistant Staphylococcus Aureus Enterocolitis
Brief Title: Biotherapy for MRSA Enterocolitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, weiyao, Institute of General Surgery, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRSA-FMT
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FMT treatment (Other): Treat the patients by fecal microbiota transplantation
  Interventions: Other: Fecal microbiota transplantation

INTERVENTIONS:
Other: Fecal microbiota transplantation — bacteria liquid from 60g fecal was infusion via nasointestinal tube for three days

SUMMARY:
Methicillin-resistant Staphylococcus aureus (MRSA) is one of the major sources of nosocomial infection. Along with the widely application of antibiotics around perioperative period, MRSA infection is increasing by years.Fecal microbial transplantation (FMT),infusion of fecal preparation from a healthy donor into the GI tract of a patient is being proposed as a novel therapeutic approach to modulate diseases associated with pathological imbalances within the resident microbiota, termed dysbiosis.It has been used to treat intestinal disease such as inflammatory bowel diseases and Clostridium difficile infection, but no reports are available on its role in treating MRSA enteritis yet. vancomycin is the first choice to treat MRSA but can also lead to an increase in antibiotic resistant organisms such as vancomycin-resistant enterococci, methicillin-resistant Staphylococcus aureus and transfer of antibiotic resistance genes among the microbial community. So FMT seems a more harmless and reasonable measure to treat similar diseases.

DETAILED DESCRIPTION:
Five cases from July, 2013 to February, 2014 were collected in Jinling hospital.They developed unexplained high fever, bloating, nausea, vomit, a high stoma output or diarrhea in the color of yellow-green with copious amounts of mucus leading to dehydration and tachycardia after short time of operation (2-4d).We got the etiology diagnosis from all the patients' gastric juice cultures which revealed MRSA.Vancocin cp had a dissatisfied effect,so FMT was supplied for treating MRSA.All the patients had a decreased intestinal flora species before FMT and the content of staphylococcus aureus almost reached half of total intestinal flora . Patients' gut bacteria after FMT gradually agree with the donors' reflected the alleviative symptoms.

ELIGIBILITY:
Inclusion Criteria:

1.18-70 years old 2.patients diagnosed as MRSA enterocolitis

Exclusion Criteria:

1.infectious diarrhea caused by other pathogenic bacteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Species diversity in fecal | one month after FMT

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Study Director — Institute of General Surgery, Jinling Hospital, Medical School of Nanjing University，
Locations (1):
- Department of General Surgery, Jinling hosptal,Medical School of Nanjing University, Nanjing, Jiangsu, China